CLINICAL TRIAL: NCT01979042
Title: Can Modern Urinary Markers be Used as Markers for Acute Kidney Failure Due to Stone Obstruction
Brief Title: Urinary Markers for Unilateral Kidney Obstruction
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CMC-12-0150-CTIL
Record Dates: First submitted 2013-10-21; First posted 2013-11-08 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Renal Colic; Acute Renal Failure
Keywords: renal colic; acute renal failure; Neutrophil gelatinase associated lipocalin
MeSH Terms: conditions — Renal Colic; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- patients with stones: 80 men and women with a normal creatinine for the past year that present in the ER with renal colic and a stone in their ureter according to imaging
- patients without stones: 20 men and women that presented in our department for elective surgery that is not related to stones or bladder outlet obstruction

SUMMARY:
Renal colic is usually caused from an obstructing stone along the ureter. Some of the patients present with a high level of creatinin in the blood, even though there is a normal functioning contralateral kidney. Furthermore creatinin is not an ideal marker for renal function during acute changes.

Several works have shown that modern urinary markers such as NGAL (neutrophil gelatinase-associated lipocalin), KIM-1 (Kidney Injury Molecule-1) and others rise earlier and are much more sensitive for kidney insult. There is a lack of research on their role in acute kidney obstruction

DETAILED DESCRIPTION:
The study population will include 100 men and women that will be recruited during the upcoming year, with a follow up of up to 3 months.

The study population will be divided into 2 groups:

1. The stone group: about 80 patients, aged 18-65, with normal creatinine for the past year that presented in our ER because of renal colic, and their imaging shows a ureteral stone.
2. The non-stone group: about 20 patients that present in our department for elective surgery not related to stones or bladder outlet obstruction.

The stone group:

---------------- In the ER the patients will be examined, undergo blood and urine workup and imaging as usual. If they are applicable according to our inclusion and exclusion criteria and admitted and they will be included in our stone group. After signing an informed consent, either as patients with a ureteral stone and normal creatinine or as patients with a ureteral stone and an abnormal creatinine, Their urine sample will be sent for the urinary markers: NGAL, KIM-1, ENdothelin and Cystatin C.

At this point it will be decided to admit or discharge them according to their clinical imaging and laboratory findings, as acceptable. The admitted patients will be followed for 48 with additional blood and urine tests.

The admitted patients that will undergo renal drainage will be a specific subgroup in which a selective urine test will be taken from the drained kidney

The non stone group:

-------------------- These are our control group from which we will take a single blood and urine test before their elective surgery.

ELIGIBILITY:
Inclusion Criteria for stone group:

* no known kidney disease
* turned to the ER due to renal colic
* imaging demonstrates a partially or totally obstructing ureteral stone

Inclusion Criteria for non stone group:

* turned to the urology department for ambulatory surgery: hydrocelectomy, varicocelectomy, stress incontinence repair,circumcision,cystoscopy

Exclusion Criteria:

* patients with stones in the contralateral ureter
* patients who underwent renal surgery
* patients who took NSAID's (nonsteroidal antiinflammatory drugs) in the past week before presentation
* patients woth anatomical defects in the kidneys

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 men and women - 80 presented in the ER with a unilateral ureteral stone and 20 presented for ambulatory surgery not related to urinary stones or bladder outlet obstruction
Sampling Method: Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2013-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
urinary markers behavior | one week
  What is the level of the urine markers NGAL, KIM-1, ENdothelin and Cystatin C at presentation and 48 hours after presentation, in patients presenting with renal colic in the ER

SECONDARY OUTCOMES:
following the markers in patients whose kidneys were drained | one week
  What is the level of the urine markers NGAL, KIM-1, ENdothelin and Cystatin C at presentation and after 48 hours after presentation, in patients with renal colic whose kidneys were drained by a ureteral stent

CONTACTS AND LOCATIONS:
Overall Officials: Ilan B Klein, MD, Principal Investigator — Carmel Medical Center; Avi Stein, Prof., Study Director — Carmel Medical Center
Locations (1):
- Carmel Lady Davis Medical Center, Haifa, Israel